CLINICAL TRIAL: NCT06201806
Title: Effect of the Consumption of a Breakfast With and Without Sweeteners (Stevia and Sucralose) on Postprandial Glycemic Response and Appetite-Satiety Sensation in Subjects With Type 1 Diabetes: A Controlled Clinical Trial.
Brief Title: To Compare Influence of Breakfast With and Without Sweeteners on Postprandial Glycemic Response and Appetite-Satiety Sensation in Subjects With Type 1 Diabetes
Acronym: T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Sociedad Chilena de Diabetes y Endocrinología (SOCHED) (Unknown)
Responsible Party: Principal Investigator, Verónica Sambra Vásquez, Clinical Professor, University of Chile
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: Proyecto Soched N°2019-04
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Non-Nutritive Sweeteners; High-Intensity Sweeteners; Sweetening Agents* / adverse effects; Male; Female; Adult; Stevia rebaudiana; Glycemic index; Sucralose; Breakfast
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Zinostatin

STUDY DESIGN:
Intervention Model Description: The study follows FAO/WHO 2008 protocol for glycemic index in breakfasts with and without non-nutritive sweeteners. Participants prep with a similar diet, light dinner, and a 10-hour fast before the test. The experimental design, implemented three times independently for 7-14 days, employs a crossover approach with each DM1 individual serving as their own control. Interventions feature test breakfasts with or without sweeteners, providing 50g of CHO. A third intervention uses white bread as a standard for glycemic response. This design calculates the area under the curve, contrasts experimental and standard responses, and determines the glycemic index for both test breakfasts.
Who Masked: Participant
Masking Description: The participant is unaware of the assigned breakfast intervention, but they were aware of consuming white bread as the standard.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test food breakfast with NCS (Experimental): Experimental: Participants with type 1 diabetes will consume Breakfast I with a mixed sweetener of stevia and sucralose, equivalent to 30 drops (36 mg stevia + 34.8 mg sucralose). Total non-nutritive sweeteners (NNS) amount to 70.8 mg.
  Intervention: Breakfast I includes whole wheat pita bread (43 g), turkey ham (40 g), gouda cheese (18 g), semi-skimmed milk 200 cc (enhanced with 15 drops of sweetener), and natural orange juice 200 cc (with an additional 15 drops of sweetener). 15 drops for each preparation, making a total of 30 drops, providing 50 grams of available carbohydrates. Subjects administer rapid-acting insulin before breakfast based on their ratio and sensitivity.
  Interventions: Other: Test food breakfast with NCS or witout NCS
- Test food breakfast without NCS (Experimental): Experimental: Intervention involves the consumption of a breakfast without non-nutritive sweeteners (NNS).
  Intervention: Subjects with type 1 diabetes who ingest Breakfast II (without sweetener): Whole wheat pita bread (43 g), turkey ham (40 g), gouda cheese (18 g), semi-skimmed milk 200 cc, and natural orange juice 200 cc.
  Intervention includes the ingestion of 50 grams of available carbohydrates in the breakfast without NNS. Subjects will administer rapid-acting insulin before breakfast based on their ratio and sensitivity.
  Interventions: Other: Test food breakfast with NCS or witout NCS
- Reference food (Active Comparator): Intervention involves the consumption of White Bread (standard food): 86g of crustless white sandwich bread as the standard food to reach the 50g of available CHO. Subjects administer rapid-acting insulin before consumption based on their ratio and sensitivity.
  Interventions: Other: Test food breakfast with NCS or witout NCS

INTERVENTIONS:
Other: Test food breakfast with NCS or witout NCS — Study Intervention: 30 drops (70.8 mg) of a stevia and sucralose mix were chosen based on Ford et al. 2011, indicating a 48 mg sucralose concentration comparable to the sweetness of a standard diet soda, due to a lack of studies on the acute effects of combined non-nutritive sweeteners.
  Glycemic Responses (GR): Blood samples collected using Accu-Chek® Instant glucometer, with fasting samples establishing baseline glucose concentration. Test breakfast or white bread consumed within 12 to 15 minutes, followed by capillary blood sampling at various intervals. Continuous glucose monitoring with a sensor was also implemented.
  Glycemic Index (GI) Calculation: Geometric calculation of the area under the curve (AUC) for each food, excluding the baseline area. Test breakfast GI determined by expressing AUC as a percentage of the standard food AUC. Final GI value averaged across groups.

SUMMARY:
Introduction: Type 1 diabetes is a chronic autoimmune disease with multifactorial etiology, resulting in partial or complete destruction of pancreatic β cells, leading to an absolute deficit of insulin and vital dependence on exogenous insulin. Treatment for type 1 diabetes (T1D) involves externally replacing the functions of pancreatic β cells through the administration of external insulin, aiming to achieve blood glucose levels close to normal ranges. Among the factors influencing postprandial glycemic excursions is the glycemic index (GI), defined as the potential of a food's carbohydrates to raise blood glucose. Many studies to date conclude that foods with a higher glycemic index (GI) result in a greater area under the curve in postprandial glycemia.

Studies in children and adults with diabetes have reported that individuals with higher non-nutritive sweetener (NNS) consumption do not exceed the acceptable daily intake (ADI) limit in most cases. Regarding the effect of non-caloric sweetener consumption on appetite-satiety and postprandial glycemia in T1D patients, there is no available evidence.

General Objective: To compare the effect of consuming a breakfast with and without sweeteners on postprandial glycemic response and appetite-satiety sensation in subjects with type 1 diabetes.

Methodology: A prospective experimental study will be conducted with non-probabilistic convenience sampling over 2 months. Thirty-two adult volunteers with T1D using intensified insulin analog schemes or insulin pumps will be recruited. Nutritional assessment and a dietary survey will be conducted to determine the habitual consumption of non-nutritive sweeteners. Two breakfasts will be tested, one with and one without non-nutritive sweeteners (separated by 7 days). Additionally, a test with White Bread (as a standard food) will be conducted. Both the standard food and the breakfast will provide 50 g of available carbohydrates in each session. Subjects will administer rapid-acting insulin before ingestion according to their ratio and sensitivity. The glycemic index of each breakfast will be determined, and the glycemic response will be analyzed using capillary glucometry and continuous glucose monitoring, with each subject serving as their own control. Finally, appetite-satiety will be determined using a visual analog scale. One-way ANOVA and the t-student test will be used for statistical analysis. Statistical analysis will be performed using IBM SPSS Statistics v.22 (SPSS Inc., Chicago, Illinois). A p-value < 0.05 will be considered significant for each analysis.

Expected Results: It is expected that the breakfast with non-nutritive sweeteners will induce a higher postprandial glycemic response, measured as a greater area under the curve in adult T1D subjects. Furthermore, it is anticipated that after consuming the breakfast with non-nutritive sweeteners, T1D subjects will experience increased appetite and reduced satiety.

DETAILED DESCRIPTION:
Experimental Design: The protocol to be used follows the procedure recommended by FAO/WHO 2008. On the day before the test, subjects will be instructed to maintain a similar intake to their usual diet, with a preferably light dinner; intense physical activity and alcohol consumption will also be restricted. Each subject will attend with a minimum fasting period of 10 hours. The foods used in the breakfast tests are specified in Table 2, and both breakfasts provide 50g of available carbohydrates (CHO).

Glycemic Responses (GR): Blood samples will be obtained through capillary blood sampling using the Accu-Chek® Instant glucometer. Two fasting blood samples will be taken, and the average result of these values will be considered as the baseline blood glucose concentration. Immediately after this, subjects will be given the test breakfast or white bread as appropriate within a time frame of 12 to 15 minutes. After 12 or 15 minutes, capillary blood samples will be taken at 30, 45, 60, 90, 120, 150, and 180 minutes after ingestion. In addition, continuous glucose monitoring with a sensor will be performed.

Calculation of the Glycemic Index (GI): The area under the curve (AUC) will be geometrically calculated for each food using the trapezoid rule, excluding the area under the baseline. To obtain the GI of the test breakfasts, the AUC of the breakfast with or without sweeteners consumed by each subject will be expressed as a percentage of the AUC increase of the standard food consumed by the same subject. The final GI value of the test breakfast with or without sweeteners will be the average of the GIs obtained in each group.

Appetite Determination: The 10 cm Visual Analog Scale (VAS) with words anchored at each end expressing the most positive and negative ratings will be used. It will be used to evaluate the sensations of hunger, satiety, and fullness, defined as follows: Hunger: "Vital and indispensable physiological need to nourish our body," Satiety: "Feeling of satisfaction, referring to satisfying the physiological need to nourish our organism," and Fullness: "State that invites stopping eating." Additionally, desire to consume food, desire for something sweet, salty, tasty, or fatty will be assessed. The person will mark their sensation on the scale, and the distance from the left end to the marked point will be measured, allowing quantification of the sensation.

Statistical Analysis: Results will be expressed as mean ± standard deviation. One-way ANOVA will be used to compare glycemic responses and the GI value between groups. Additionally, t-student will be used to compare glycemic responses between breakfasts. Statistical analysis will be performed using the IBM SPSS Statistics v.22 statistical program (SPSS Inc., Chicago, Illinois). A p-value < 0.05 will be considered significant for each analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 1 diabetes (DM1) aged between 18 and 60 years.
* Confirmed diagnosis of DM1.
* Users of an intensified regimen with insulin analogs (multiple doses) or users of an insulin pump.

Exclusion Criteria:

* History of celiac disease.
* Allergy and/or food intolerances to any of the test foods.
* Subjects who carry out moderate to intense physical activity three or more times a week for more than 30 minutes at a time
* Subjects with the use of vitamin supplements or antioxidants
* Subjects with an allergy or aversion to the sweeteners used in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Glycemic Responses (GR) | time frame of 12 to 15 minutes. After this period, capillary blood samples were collected at 30, 45, 60, 90, 120, 150, and 180 minutes post-ingestion.
  Blood samples were collected through capillary blood sampling using the Accu-Chek® Instant glucometer. Two fasting blood samples were taken, and the average result of these values was considered as the baseline blood glucose concentration. Subsequently, participants were provided with the test breakfast or white bread, as appropriate, within a time frame of 12 to 15 minutes. After this period, capillary blood samples were collected at 30, 45, 60, 90, 120, 150, and 180 minutes post-ingestion. Additionally, continuous glucose monitoring with a sensor was conducted.

SECONDARY OUTCOMES:
Determination of Nutritional Status: | Once time in the beggining of the study
  Each participant was asked to wear light clothing and remove their shoes. Subsequently, body weight was measured using a scale with an accuracy of 0.1 kg. Height was measured in centimeters (cm) using a stadiometer with an accuracy of 0.1 cm. Nutritional status was classified according to the World Health Organization (WHO) 2000 report.
Determination of Sweetener Intake (Modified Consumption Trend Survey): | Once time in the beggining of the study
  A retrospective survey was administered, prompting participants to recall their dietary habits over a one-month period. The survey gathered information on specific food consumption patterns, emphasizing the frequency of intake of items containing added sweeteners and discretionary sweetener consumption. This assessment also aimed to identify participants categorized as high or low consumers of non-nutritive sweeteners (NNS).
Assessment of Appetite: | It is measured at the beginning of the intervention, as well as at 60 and 120 minutes after the start.
  The 10 cm Visual Analog Scale (VAS) with anchored words at each end was employed. This scale expresses the most positive and negative ratings. It was utilized to evaluate the sensations of hunger, satiety, and fullness, defined as follows: Hunger: "Vital and indispensable physiological need to nourish our body," Satiety: "Feeling of satisfaction, related to fulfilling the physiological need to nourish our body," and Fullness: "State that encourages stopping eating." Additionally, desires for consuming specific foods, such as something sweet, salty, tasty, or fatty, were included. Participants marked their sensations on the scale, and the distance from the left end to the marked point was measured, allowing for the quantification of the sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chile. Faculty of Medicine, Santiago, Chile